CLINICAL TRIAL: NCT02240108
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Multiregional, One Year Study to Assess the Efficacy and Safety of Twice Daily Oral Rifaximin Delayed Release Tablets for Induction of Clinical Remission With Endoscopic Response at 16 Weeks Followed by Clinical and Endoscopic Remission at 52 Weeks in Subjects With Active Moderate Crohn's Disease
Brief Title: One Year Study of Rifaximin Delayed Release (DR) in Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to difficulty in enrollment and lack of clinical study drug access.
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Salix Pharmaceuticals, Inc. a division of Bausch Health US, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECD3126
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Rifaximin; Clinical remission with endoscopic response; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin EIR 800 mg (Experimental): Participants will receive rifaximin EIR 400 milligrams (mg) tablets orally twice daily for 52 weeks.
  Interventions: Drug: Rifaximin EIR
- Placebo (Placebo Comparator): Participants will receive placebo matching to rifaximin EIR tablets orally twice daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin EIR — Rifaximin EIR tablets will be administered per the dose and schedule specified in the arm.
  Arms: Rifaximin EIR 800 mg
Drug: Placebo — Placebo matching to rifaximin EIR tablets will be administered per the dose and schedule specified in the arm.
  Arms: Placebo

SUMMARY:
The primary objective is to determine the efficacy of rifaximin DR also referred to as Extended Intestinal Release (EIR) tablets vs. placebo for the induction of clinical remission and endoscopic response following 16 weeks of treatment in participants presenting with active moderate Crohn's disease. A key secondary objective is to evaluate clinical and endoscopic remission following an additional 36 weeks of treatment.

DETAILED DESCRIPTION:
RECD3126 is a double-blind, placebo-controlled, parallel-group, multicenter, multiregional, 52-week study to assess the efficacy and safety of rifaximin DR tablets for the induction of clinical remission and endoscopic response at 16 weeks followed by clinical and endoscopic remission after 52 weeks of continuous therapy in participants with active moderate Crohn's disease.

Participants will be randomized in a 1:1 allocation to rifaximin or placebo at the beginning of the treatment period and will maintain treatment assignment throughout the duration of the study. Ileocolonoscopy will be performed on all participants at baseline, between Weeks 16 and 17 (end of the Induction Phase), and following completion of the 36-week Long Term Treatment Phase (Week 52).

ELIGIBILITY:
Major Inclusion Criteria:

* Moderate, non-fistulizing Crohn's disease in the ileum and/or colon prior to randomization; and a SES-CD score of ≥7 (confirmed by centralized endoscopy reading).
* During the screening period, the participant will need to have certain average daily scores for abdominal pain and average number of liquid/very soft stools.

Major Exclusion Criteria:

* Pregnant or lactating females. Females of childbearing (reproductive) potential must have a negative serum pregnancy test at screening and agree to use a highly effective method(s) of contraception throughout their participation in the study. Diagnosis of ulcerative or indeterminate colitis.
* Diagnosis of Celiac Disease.
* Bowel surgery within 12 weeks prior to screening and/or has surgery planned or deemed likely for Crohn's disease during the study period.
* Presence of an ileostomy or colostomy.
* Known fixed symptomatic stenosis/stricture of the small or large bowel.
* Had more than one segmental colonic resection.
* Had more than 3 small bowel resections or symptoms associated with short bowel syndrome.
* Current evidence of peritonitis.
* History or evidence of colonic mucosal dysplasia.
* History or evidence of adenomatous colonic polyps that have not been removed.
* Unwilling to be tapered off corticosteroids by Week 8 or the participant is known by the Investigator to be steroid-dependent.
* Has used a biologic within 12 weeks of randomization.
* Used cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, or similar drugs within 8 weeks prior to randomization.
* Had rectal administration of 5-aminosalicylic acid (5-ASA) or corticosteroid enemas/foams/ suppositories within 2 weeks prior to screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (71):
- United States (71):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Sherwood, Arkansas
  - Garden Grove, California
  - La Jolla, California
  - La Mirada, California
  - Laguna Hills, California
  - Los Angeles, California
  - Northridge, California
  - Oceanside, California
  - San Diego, California
  - Littleton, Colorado
  - Waterbury, Connecticut
  - Boca Raton, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Hollywood, Florida
  - Inverness, Florida
  - Lauderdale Lakes, Florida
  - Maitland, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - Iowa City, Iowa
  - Crestview Hills, Kentucky
  - Shreveport, Louisiana
  - West Monroe, Louisiana
  - Hagerstown, Maryland
  - Hollywood, Maryland
  - Brockton, Massachusetts
  - Caro, Michigan
  - Stevensville, Michigan
  - Wyoming, Michigan
  - Plymouth, Minnesota
  - Ocean Springs, Mississippi
  - Tupelo, Mississippi
  - Bridgeton, Missouri
  - Creve Coeur, Missouri
  - Vineland, New Jersey
  - Voorhees Township, New Jersey
  - New York, New York
  - Fayetteville, North Carolina
  - Kinston, North Carolina
  - Beavercreek, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Lima, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Columbia, South Carolina
  - Fort Mill, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Humble, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Ogden, Utah
  - West Jordan, Utah
  - West Valley City, Utah
  - Chesapeake, Virginia
  - Richland, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 81 participants were enrolled and randomized in this study.
Pre-assignment Details: Participants were randomized in a 1:1 allocation to Rifaximin EIR 800 mg or Placebo at the beginning of the treatment period and were maintained on that treatment assignment for 16 weeks, followed by an open-label long-term active treatment extension of an additional 36 weeks.
Groups:
- Rifaximin EIR 800 mg: Participants received rifaximin extended intestinal release (EIR) 400 milligrams (mg) tablets orally twice daily for 52 weeks.
- Placebo: Participants received placebo matched to rifaximin EIR tablets orally twice daily for 52 weeks.
Period: Overall Study
Arm/Group | Rifaximin EIR 800 mg | Placebo
Started | 35 | 46
Intent-to-treat (ITT) Population (Received at least 1 dose of study drug) | 35 | 45
Completed | 21 | 21
Not Completed | 14 | 25
Not completed — Other than specified | 8 | 6
Not completed — Adverse Event | 1 | 9
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 4 | 9
Not completed — StudyTerminated by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who took at least 1 dose of study drug.
Groups:
- Rifaximin EIR 800 mg: Participants received rifaximin EIR 400 mg tablets orally twice daily for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Rifaximin EIR 800 mg | Placebo | Total
Number analyzed (Participants) | 35 | 45 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.85) | 43.2 (12.97) | 43.3 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 16 | 21 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 31 | 38 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 29 | 38 | 67
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Crohn's Disease Activity Index (CDAI) Score [Mean (Standard Deviation); unit: units on a scale] — CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
  units on a scale | 305.4 (69.51) | 300.0 (56.39) | 302.4 (62.11)
Simple Endoscopic Score for Crohn's Disease (SES-CD) [Mean (Standard Deviation); unit: units on a scale] — SES-CD is a validated instrument reflecting an endoscopist's global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. The total SES-CD was calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease.
  units on a scale | 12.0 (5.01) | 11.7 (4.61) | 11.8 (4.76)
Duration of Disease [Mean (Standard Deviation); unit: years] — Duration of Crohn's disease at baseline was measured.
  years | 10.5 (8.57) | 9.6 (9.53) | 10.0 (9.08)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 1) at Week 16
Description: Clinical symptom remission defined by (1) the total number of liquid/very soft stools for the 7 days prior to the Week 16 visit being less than or equal to (≤) 10 (from CDAI Item 1). CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 16
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 6 | 8

2. Primary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 2) at Week 16
Description: Clinical Symptom Remission defined by (2) an abdominal pain (graded from 0 [less severe]-3 [more severe]) rating of ≤ 1 (from CDAI Item 2) on each day for the 7 days prior to the Week 16 visit. CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 16
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 19 | 15

3. Primary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 1 and 2 Both) at Week 16
Description: Clinical Symptom Remission defined by (1) the total number of liquid/very soft stools for the 7 days prior to the Week 16 visit being ≤ 10 (from CDAI Item 1); and (2) an abdominal pain (graded from 0 [less severe]-3 [more severe]) rating of ≤ 1 (from CDAI Item 2) on each day for the 7 days prior to the Week 16 visit. CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 16
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 5 | 7

4. Primary Outcome: Number of Participants With Endoscopic Response Between Week 16 and 17
Description: Endoscopic response defined as a ≥ 3-point decrease in the SES-CD from baseline to the SES-CD score obtained between Week 16 and Week 17. SES-CD scores were calculated from centrally-read digital video of ileocolonoscopies performed at baseline and between Week 16 and Week 17. SES-CD is a validated instrument reflecting an endoscopist's global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. The total SES-CD was calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 16 to 17
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 10 | 10

5. Primary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 1) at Week 52
Description: Clinical symptom remission defined by (1) the total number of liquid/very soft stools for the 7 days prior to the Week 52 visit being ≤ 10 (from CDAI Item 1). CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 52
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 7 | 3

6. Primary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 2) at Week 52
Description: Clinical Symptom Remission defined by (2) an abdominal pain (graded from 0 [less severe]-3 [more severe]) rating of ≤ 1 (from CDAI Item 2) on each day for the 7 days prior to the Week 52 visit. CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 52
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 9 | 5

7. Primary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 1 and 2 Both) at Week 52
Description: Clinical Symptom Remission defined by (1) the total number of liquid/very soft stools for the 7 days prior to the Week 52 visit being ≤ 10 (from CDAI Item 1); and (2) an abdominal pain (graded from 0 [less severe]-3 [more severe]) rating of ≤ 1 (from CDAI Item 2) on each day for the 7 days prior to the Week 52 visit. CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 52
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 6 | 1

8. Primary Outcome: Number of Participants With Endoscopic Response at Week 52
Description: Endoscopic response defined as a ≥ 3-point decrease in the SES-CD from baseline to the SES-CD score obtained at Week 52. SES-CD is a validated instrument reflecting an endoscopist's global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. The total SES-CD was calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 52
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 9 | 15

9. Secondary Outcome: Number of Participants Who Achieved Clinical Remission (Defined as CDAI Score of <150) at Week 16
Description: Clinical remission was defined as a CDAI score of less than 150 points at Week 16. CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: Week 16
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 17 | 12

10. Secondary Outcome: Number of Participants Who Achieved Clinical Symptom Remission (From CDAI Item 1 and 2 Both) Over Time
Description: Clinical Symptom Remission defined by (1) the total number of liquid/very soft stools for the 7 days prior to each clinical visit being ≤ 10 (from CDAI Item 1); and (2) an abdominal pain (graded from 0 [less severe]-3 [more severe]) rating of ≤ 1 (from CDAI Item 2) on each day for the last 7 days prior to each clinic visit in ≥ 80% of the study visits during the 52-week treatment period, including Week 52. CDAI score is a weighted, composite index of 8 items (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extraintestinal manifestations including fistula, use or non-use of antidiarrheal agents, presence or absence of abdominal mass, hematocrit, and body weight). Scores range from 0 to approximately 600 with higher scores indicating greater disease severity.
Time Frame: From Baseline to Week 52
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 2 | 3

11. Secondary Outcome: Number of Participants With SES-CD Score of 0 at Week 52
Description: SES-CD is a validated instrument reflecting an endoscopist's global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. The total SES-CD was calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease.
Time Frame: Week 52
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin EIR 800 mg | Placebo
Number analyzed (Participants) | 35 | 45
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from time of signing informed consent until the end of the follow-up period (2 weeks after last treatment [Week 54]) .
Description: Occurrences of AEs or serious adverse events (SAEs) were reported during each study visit or by the participant outside of scheduled visits.
Arm/Group | Rifaximin EIR 800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/45
Serious Adverse Events (participants affected / at risk) | 6/35 | 9/45
Other Adverse Events (participants affected / at risk) | 25/35 | 25/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin EIR 800 mg (N=35) | Placebo (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin EIR 800 mg (N=35) | Placebo (N=45)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Crohn's disease (Gastrointestinal disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 3 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4
Fatigue (General disorders) | 2 | 2
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1
Pharyngitis streptococcal (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulty in enrollment and lack of clinical study drug access. The efficacy results are not considered definitive and are considered for exploratory purposes only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (2):
  • Study Protocol (2014-07-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02240108/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT02240108/SAP_001.pdf